CLINICAL TRIAL: NCT07381855
Title: Biosignatures for the Development of Attention Deficit Hyperactivity Disorder
Acronym: AHEAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-14-0158-CR11; R01MH112588 (NIH)
Record Dates: First submitted 2026-01-20; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: ADHD; Disruptive Behaviours
Keywords: ADHD; callous-unemotional behaviors; summer treatment program; young children; school readiness; emotion dysregulation; parenting
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Summer Treatment Program for children transitioning to and from kindergarten (STP-K) (Experimental): Participants in the STP-K included children ages 4 to 7 who attended a school readiness class during the summer, Monday-Friday from 8 a..m to 4:00 p.m. for 7 to 8 weeks.
  Parents received feedback everyday in the form of daily report card regarding how their children performed during the day.
  Parents also attended a weekly parenting program lasting between 1.5 to 2 hours.
  Interventions: Behavioral: Summer treatment program for children transitioning to and from kindergarten (STP-K)

INTERVENTIONS:
Behavioral: Summer treatment program for children transitioning to and from kindergarten (STP-K) — The STP-K is a multimodal intervention including a school readiness class, which consists of a behavior modification program as well as an academic and social-emotional curriculum, along with a parenting program.
  Throughout the day children participate in activities designed to promote a) behavioral and social-emotional skills consistent with the expectations of kindergarten and first grade, b) academic skills, c) physical activity, good sportsmanship, basic sports skills, and c) a positive attitude towards learning and school. Fifteen children are assigned to a classroom, staffed by one lead teacher, one lead counselor, and four paraprofessional developmental aides, yielding a 2:5 staff to student ratio. A behavior modification program is used across activities to promote positive behaviors.
  Parents then receive feedback everyday on how their child is doing and also attend a weekly parenting program lasting between 1.5 to 2 hours.
  Other Names: Summer Treatment Program; Summer Treatment Program for Prekindergarteners (STP-PreK)

SUMMARY:
As an exploratory aim of this grant, we examined the extent to which a comprehensive psychosocial intervention conducted in the summer can improve young children with disruptive behavior challenges as it relates to their social-emotional and academic functioning.

DETAILED DESCRIPTION:
Due to the high prevalence rates and significant impairments associated with ADHD and comorbid disruptive behavior disorders, it is not surprising that a great deal of research has focused on psychosocial interventions, with the Summer Treatment Program (STP) emerging as one of the most widely regarded and effective multimodal psychosocial treatments for children with ADHD and comorbid disruptive behavior disorders. Over the last 15 years, the STP has been adapted for preschoolers transitioning into kindergarten, with similar success in not only improving general externalizing behavior problems (EBP), but also other school readiness outcomes.

Part of the STP for pre-kindergarteners' (STP-PreK) successful adaption is due to the recognition of the importance of addressing children's emotion dysregulation, which has not only been identified as a core impairment among children with ADHD but also a contributing factor in the development of DBDs. Callous-unemotional traits (CU) is one emotion dysregulation domain that amplifies impairments associated with ADHD and DBDs, and can attenuate the response to evidence-based treatments. The current study examines the extent to which the STP-PreK can improve these emotion dysregulation outcomes along with other school readiness outcomes (i.e., academic functioning and social skills) in a sample of young children with ADHD and co-occurring DBDs, compared to their TD peers.

ELIGIBILITY:
Inclusion Criteria:

* Children had to be attending school and between the ages of 4 and 7
* Children in the typically developing (TD) group had to have their parents and/or their teachers endorse them as having less than four ADHD symptoms (across either Inattention or Hyperactivity/Impulsivity), less than four ODD symptoms, less than three CD symptoms, and indicated no clinically significant impairment (score below 3 on the IRS).
* Children in the ADHD group had to have endorsed at least 6 ADHD symptoms of Inattention and/or Hyperactivity/Impulsivity, land indicated clinically significant impairment (score above 3 on the IRS) across parent and/or teacher report.
* Children in the ADHD group also had to attend the STP-K.

Exclusion Criteria:

* Diagnosis of Autism Spectrum Disorder
* Full scale IQ below 70
* Currently taking any psychotropic medication

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 323 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Overall Emotion Regulation as measured by the Emotion Regulation Checklist | Baseline
  The average score on the emotion regulation subscale of the 24-item Emotion Regulation Checklist was used with higher scores indicating better emotion regulation skills.
Overall Emotion Regulation as measures by the Emotion regulation Checklist | 6 months after enrollment (post treatment)
  The average score on the emotion regulation subscale of the 24-item Emotion Regulation Checklist was used with higher scores indicating better emotion regulation skills.
Overall Emotion Regulation as measured by the Emotion regulation Checklist | 1 year after enrollment
  The average score on the emotion regulation subscale of the 24-item Emotion Regulation Checklist was used with higher scores indicating better emotion regulation skills.
ADHD symptoms as assesed by the Disruptive Behavior Disorders Rating Scale | Baseline
  Average symptom severity of the ADHD items of the Disruptive Behavior Disorders Rating Scale with higher scores indicating worse ADHD severity.
ADHD symptoms as assessed by the Disruptive Behavior Disorders Rating Scale | 6 months after enrollment (post-treatment)
  Average symptom severity of the ADHD items of the Disruptive Behavior Disorders Rating Scale with higher scores indicating worse ADHD severity.
ADHD symptoms as assessed by the Disruptive Behavior Disorders Rating Scale | Completed 1 year after enrollment
  Average symptom severity of the ADHD items of the Disruptive Behavior Disorders Rating Scale with higher scores indicating worse ADHD severity.
Overall Adaptive Functioning as assessed by the Behavior Assessment System for Children | baseline
  T-score on the adaptive functioning subscale of the Behavior Assessment System for Children with higher scores indicating better adaptive functioning skills
Overall adaptive functioning as measured by the Behavior Assessment System for Children | 6 months after enrollment (post-treatment)
  T-score on the adaptive functioning subscale of the Behavior Assessment System for Children with higher scores indicating better adaptive functionining skills
Overall adaptive functioning as assessed by the Behavior Assessment System for Children | Completed 1 year after enrollment
  t-score on the adaptive functioning subscale of the Behavior Assessment System for Children with higher scores indicating better adaptive functionining skills
Severity of Disruptive Behaviors as assessed by the Disruptive Behavior Disorders Rating Scale | baseline
  Average symptom severity of the ODD and CDD items of the Disruptive Behavior Disorders Rating Scale with higher scores indicating worse disruptive behaviors.
Severity of Disruptive behaviors as assessed by the Disruptive Behavior Disorders Rating Scale | 6 months after enrollment (post-treatment)
  Average symptom severity of the ODD and CDD items of the Disruptive Behavior Disorders Rating Scale with higher scores indicating worse disruptive behaviors.
Severity of Disruptive Behaviors as assessed by the Disruptive Behavior Disorders Rating Scale | 1 year after enrollment
  Average symptom severity of the ODD and CDD items of the Disruptive Behavior Disorders Rating Scale with higher scores indicating worse disruptive behaviors.
Severity of callous-unemotional behaviors as assessed by the abbreviated version of the Inventory of Callous-Unemotional Traits. | baseline
  Average frequency of callous-unemotional behaviors across the 12 items of the questionnaire with higher scores indicating more severe behaviors.
Severity of callous-unemotional behaviors as assessed by the abbreviated version of the Inventory of Callous-Unemotional Traits | 6 months after enrollment (post-treatment)
  Average frequency of callous-unemotional behaviors across the 12 items of the questionnaire with higher scores indicating more severe behaviors.
Severity of callous-unemotional behaviors as assessed by the abbreviated version of the Inventory of Callous-unemotional traits. | 1 year after enrollment
  Average frequency of callous-unemotional behaviors across the 12 items of the questionnaire with higher scores indicating more severe behaviors.
Social Skills as assessed via the Behavior Assessment System for Children | baseline
  T-score on the social skills subtest of the Behavior Assessment System for Children with higher scores indicating better social skills.
Social Skills as assessed by the Behavior Assessment System for Children | 6 months after enrollment (post-treatment)
  T-score on the social skills subtest of the Behavior Assessment System for Children with higher scores indicating better social skills.
Social Skills as assessed by the Behavior Assessment System for Children | 1 year after enrollment
  T-test on the social skills subtest of the Behavior Assessment System for Children with higher scores indicating better social skills
Overall social problem solving as assessed by the Challenging Situations Task | baseline
  Total prosocial score across the six hypothetical peer situations from the Challenging Situations task with higher scores indicating better social-problem solving.
Overall social problem solving as assessed by the Challenging Situations Task | 6 months after enrollment (post-treatment)
  Total prosocial score across the six hypothetical peer situations from the Challenging Situations task with higher scores indicating better social-problem solving.
Overall social problem solving as assessed by the Challenging Situations Task | 1 year after enrollment
  Total prosocial score across the six hypothetical peer situations from the Challenging Situations task with higher scores indicating better social-problem solving.
Overall Academic Achievement as measured by the Woodcock Johnson Test of Achievement | baseline
  The current study examined the mean raw scores of the derived composite scores on the Woodcock-Johnson Test of Achievement: Brief Reading (letter-word identification, passage comprehension), Brief Math (applied problems, calculation), and Brief Writing (spelling, writing samples). However, given the high correlations among these composites, an overall achievement composite was used with higher scores indicating better academic functioning.
Overall Academic Achievement as measured by the Woodcock Johnson Test of Achievement | 6-months after enrollment (post-treatment)
  The current study examined the mean raw scores of the derived composite scores on the Woodcock-Johnson Test of Achievement: Brief Reading (letter-word identification, passage comprehension), Brief Math (applied problems, calculation), and Brief Writing (spelling, writing samples). However, given the high correlations among these composites, an overall achievement composite was used with higher scores indicating better academic functioning.
Overall Academic Achievement as measured by the Woodcock Johnson Test of Achievement | 1 year after enrollment
  The current study examined the mean raw scores of the derived composite scores on the Woodcock-Johnson Test of Achievement: Brief Reading (letter-word identification, passage comprehension), Brief Math (applied problems, calculation), and Brief Writing (spelling, writing samples). However, given the high correlations among these composites, an overall achievement composite was used with higher scores indicating better academic functioning.
Overall readiness for kindergarten as assessed by the Kindergarten Behavior and Academic Competency Scale | baseline
  An overall score from the 23-items of the Kindergarten Behavior and Academic Competency Scale, which measures kindergarten readiness across domains (following clasroom rules, completing academic work) was derived by averaging across all items (along a 5-point scale) with higher scores indicating greater kindergarten readiness
Overall readiness for kindergarten as assessed by the Kindergarten Behavior and Academic Competency Scale | 6 months after enrollment
  An overall score from the 23-items of the Kindergarten Behavior and Academic Competency Scale, which measures kindergarten readiness across domains (following clasroom rules, completing academic work) was derived by averaging across all items (along a 5-point scale) with higher scores indicating greater kindergarten readiness
Overall readiness for kindergarten as assessed by the Kindergarten Behavior and Academic Competency Scale | 1 year after enrollment
  An overall score from the 23-items of the Kindergarten Behavior and Academic Competency Scale, which measures kindergarten readiness across domains (following clasroom rules, completing academic work) was derived by averaging across all items (along a 5-point scale) with higher scores indicating greater kindergarten readiness
Overall academic readiness for kindergarten as assessed by the Bracken School Readiness Assessment | baseline
  The Bracken School Readiness Assessment is a widely-used and psychometrically sound test consisting of five subtests assessing children's receptive knowledge of colors, letters, numbers/counting, sizes/comparisons, and shapes. For this study, the overall school readiness composite raw score was used with higher scores indicating better academic skills.
Overall academic readiness for kindergarten as assessed by the Bracken School Readiness Assessment | Completed 6 months after enrollment
  The Bracken School Readiness Assessment is a widely-used and psychometrically sound test consisting of five subtests assessing children's receptive knowledge of colors, letters, numbers/counting, sizes/comparisons, and shapes. For this study, the overall school readiness composite raw score was used with higher scores indicating better academic skills.
Overall academic readiness for kindergarten as assessed by the Bracken School Readiness Assessment | Completed 1 year after enrollment
  The Bracken School Readiness Assessment is a widely-used and psychometrically sound test consisting of five subtests assessing children's receptive knowledge of colors, letters, numbers/counting, sizes/comparisons, and shapes. For this study, the overall school readiness composite raw score was used with higher scores indicating better academic skills.
Observed Emotion Regulation as assessed via the Laboratory Temperament Assessment Battery | baseline
  A global measure of emotion regulation was coded (on a scale of 0 to 4) from two frustration tasks from the Laboratory Temperament Assessment Battery with higher average scores indicating better emotion regulation skills.
Observed Emotion Regulation as assessed via the Laboratory Temperament Assessment Battery | 6 months after enrollment (post treatment)
  A global measure of emotion regulation was coded (on a scale of 0 to 4) from two frustration tasks from the Laboratory Temperament Assessment Battery with higher average scores indicating better emotion regulation skills.
Observed Emotion Regulation as assessed via the Laboratory Temperament Assessment Battery | 1 year after enrollment
  A global measure of emotion regulation was coded (on a scale of 0 to 4) from two frustration tasks from the Laboratory Temperament Assessment Battery with higher average scores indicating better emotion regulation skills.
Overall Executive functioning as measured by the Behavior Rating Inventory of Executive Function | baseline
  T-score of the emergent metacognitive index of the Behavior Rating Inventory of Executive Function was used (items are rated on a three point liker scale) with higher scores indicating poorer executive functioning
Overall Executive functioning as measured by the Behavior Rating Inventory of Executive Function | 6 months after enrollment
  T-score of the emergent metacognitive index of the Behavior Rating Inventory of Executive Function was used (items are rated on a three point liker scale) with higher scores indicating poorer executive functioning
Overall Executive functioning as measured by the Behavior Rating Inventory of Executive Function | 1 year after enrollment
  T-score of the emergent metacognitive index of the Behavior Rating Inventory of Executive Function was used (items are rated on a three point liker scale) with higher scores indicating poorer executive functioning
Overall Executive Functioning Performance as measured by the Head-Toes-Knees-Shoulders task | baseline
  Total score on the Head-Toes-Knees-Shoulders task, which consists of 10 test trials. Scores range from 0 to 40 with higher scores indicative of better executive functioning.
Overall Executive Functioning Performance as measured by the Head-Toes-Knees-Shoulders task | 6 months after enrollment
  Total score on the Head-Toes-Knees-Shoulders task, which consists of 10 test trials. Scores range from 0 to 40 with higher scores indicative of better executive functioning.
Overall Executive Functioning Performance as measured by the Head-Toes-Knees-Shoulders task | 1 year after enrollment
  Total score on the Head-Toes-Knees-Shoulders task, which consists of 10 test trials. Scores range from 0 to 40 with higher scores indicative of better executive functioning.
Peer status as assessed by sociometrics ratings during the intervention | Through study completion, an average of 1 year
  A Social Preference Index score capturing overall peer status within the classroom was derived by subtracting the child's "like least" nominations from their peers from their standardized "like most" nominations from their peers, then re-standardized, as is commonly done in sociometric analyses. Higher social preference scores indicate higher peer status relative to other children in their class.

SECONDARY OUTCOMES:
Intervetion Attendance | Through study completion, an average of 1 year
  As part of the intervention (STP-K), children attend the summer camp and parents attend weekly parent training. The overall number of days attended will be used with higher numbers indicating greater participation in the intervention.
Daily Report Card | Through study completion, an average of 1 year
  Children's daily report card performance defined by percentage of days in which their behavior and academic goals were achieved leading to a "green" (75% or better) "yellow (50-74%)" or "red (below 50%)" day across the STP-K.

IPD SHARING:
Plan to Share IPD: No
We already have our data in the National Institute of Mental Health Data Archive (NDA)